CLINICAL TRIAL: NCT03109184
Title: Partner Violence Prevention for Middle School Boys: A Dyadic Web-Based Intervention
Brief Title: Violence Prevention for Middle School Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 504616
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-03

CONDITIONS: Intimate Partner Violence
Keywords: Dating violence prevention; Adolescent boys; Middle school; Web-based prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (No Intervention): Parents and teens enrolled in the study and randomized to the control condition wait until they complete their 3-month and 9-month follow-up surveys before completing the web-based program.
- Project STRONG (Experimental): The web-based program consists of a number of games, activities, and didactic information that teens move through with their parent. Didactic information introduces teens and parents to specific emotion management, communication, and problem solving strategies as well as sexual health and healthy relationship information. Games and activities allow parents and teens to practice and apply strategies to developmentally appropriate situations.
  Interventions: Behavioral: Project STRONG

INTERVENTIONS:
Behavioral: Project STRONG — The web-based program consists of a number of games, activities, and didactic information that teens move through with their parent. Didactic information introduces teens and parents to specific emotion management, communication, and problem solving strategies as well as sexual health and healthy relationship information. Games and activities allow parents and teens to practice and apply strategies to developmentally appropriate situations.
  Arms: Project STRONG

SUMMARY:
This study will develop and test a web-based intervention to enhance emotion regulation skills and parent-son relationship communication to decrease adolescent boys' risk for dating violence involvement as well as attitudes supporting relationship aggression.

DETAILED DESCRIPTION:
Over the past ten years dating violence (DV) has been recognized as a significant public health problem affecting adolescents. Emerging data suggest that boys and girls have different developmental trajectories toward violence and therefore prevention programs that target their unique pathways to DV are needed. Despite this need, there is a relative dearth of such gender-informed programs for early adolescent boys. This research project aims to prevent the emergence of DV perpetration/ victimization among boys by developing a web-based intervention that is informed by research on gender-specific pathways to violence and harnesses the influence of parents during the early adolescent years.

Among boys, the perpetration of delinquency-related violence and attitudes supporting violence has been found to predict later perpetration of DV. Thus, gender-informed interventions designed to prevent DV in boys need to target skills that underlie violent behavior and attitudes. The goal of this study is to develop and test a web-based intervention to enhance emotion regulation skills and parent-son relationship communication to prevent DV.

Development and testing will occur in three phases. In the Development Phase, the intervention modules will be developed and iteratively reviewed by both a panel of experts familiar with the research in the field as well as an advisory group of parents and teens from the target population. In the Acceptability Testing Phase, testing will be conducted to assess acceptability and feasibility, and this will be followed by revisions to the intervention program based on feedback and observations. During the Randomized Controlled Trial (RCT) Phase, 120 families will complete the intervention program in an observed setting, to ensure fidelity to intervention dosing. Parents and adolescents will complete the program together and then complete assessments of aggressive and risk behaviors, parent-child communication, and emotion regulation at baseline, 3-,and 9-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 1) adolescent enrolled in the 7th or 8th grade,
* 2) parent/legal guardian and teen are English speaking,
* 3) parent/legal guardian is willing to provide consent for the adolescent to participate in the study,
* 4) adolescent is willing to provide assent for their own participation.

Exclusion Criteria:

* 1) observable cognitive or developmental delays that would preclude participation,
* 2) residing with participating parent/guardian less than half time

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Eligibility based on youth self-representation as male gender
Enrollment: 119 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christie Rizzo, PhD, Principal Investigator — Northeastern University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizzo CJ, Houck C, Barker D, Collibee C, Hood E, Bala K. Project STRONG: an Online, Parent-Son Intervention for the Prevention of Dating Violence among Early Adolescent Boys. Prev Sci. 2021 Feb;22(2):193-204. doi: 10.1007/s11121-020-01168-6. Epub 2020 Sep 17. PMID 32940857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were individually randomized at the level of the dyad, thus our study randomized 119 dyads. Parents and teens were not randomized separately. There were only two study arms, CONTROL families and STRONG families.
Period: Overall Study
Arm/Group | Waitlist Control | Project STRONG
Started | 60 | 59
Completed | 53 | 52
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: A completer analysis was deemed appropriate as the small sample size of this pilot study could be impacted substantially from inadequate intervention dose. Analyses included intervention families who received an adequate dose of intervention, defined as a minimum of 4 out of 6 intervention modules (n=114/119).
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control | Project STRONG | Total
Number analyzed (Participants) | 60 | 54 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] — Teen Report
  years | 13.05 (0.7) | 13.04 (0.7) | 13.04 (0.7)
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent Report
  years | 42.52 (7.18) | 42.54 (6.31) | 42.53 (6.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Teen Report
  Participants
    Female | 0 | 0 | 0
    Male | 60 | 54 | 114
Sex: Female, Male [Count of Participants; unit: Participants] — Parent Report
  Participants
    Female | 54 | 48 | 102
    Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Teen Report
  Participants
    Hispanic or Latino | 12 | 15 | 27
    Not Hispanic or Latino | 48 | 39 | 87
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent Report
  Participants
    Hispanic or Latino | 10 | 11 | 21
    Not Hispanic or Latino | 46 | 41 | 87
    Unknown or Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Teen Report
  Participants
    White | 30 | 26 | 56
    Non-white | 30 | 28 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Parent Report
  Participants
    White | 43 | 38 | 81
    Non-white | 17 | 15 | 32
    Unknown/Not-reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Enrollment was by dyad
  participants
    United States | 60 | 54 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change in Dating Violence (DV) Perpetration From Baseline to 9 Months
Description: The Conflict in Adolescent Dating Relationships Inventory (CADRI) is a behavioral measure of abuse perpetration and victimization. It was completed by teens in reference to conflict or disagreement with a current or recent dating partner. Each question is asked twice, first regarding perpetration and, again in relation to victimization producing a perpetration and a victimization sub scale. Percentages include teens endorsing any perpetration or victimization.
Time Frame: Baseline, 3 months, and 9 months
Population: COMPLETER ANALYSIS
Measure: Count of Participants; unit: Participants
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
Participants
  Baseline DV Perpetration: DV Absent | 46 | 40
  Baseline DV Perpetration: DV Present | 14 | 14
  3-month DV Perpetration: DV Absent | 50 | 43
  3-month DV Perpetration: DV Present | 10 | 11
  9-month DV Perpetration: DV Absent | 49 | 45
  9-month DV Perpetration: DV Present | 11 | 9
  Baseline DV Victimization: DV Absent | 46 | 41
  Baseline DV Victimization: DV Present | 14 | 13
  3-month DV Victimization: DV Absent | 50 | 40
  3-month DV Victimization: DV Present | 10 | 14
  9-month DV Victimization: DV Absent | 50 | 43
  9-month DV Victimization: DV Present | 10 | 11
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Odds Ratio (OR) = 1.21 — 3-Month follow-up between groups odds ratio of DV perpetration
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Odds Ratio (OR) = 0.61 — 9-month follow-up between group odds ratio of DV perpetration
Statistical Analysis 3: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Odds Ratio (OR) = 1.79 — 3-month follow-up between groups odds ratio of DV victimization
Statistical Analysis 4: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Odds Ratio (OR) = 0.86 — 9-month follow-up between groups odds ratio of DV victimization

2. Primary Outcome: Change in General Aggressive Behavior From Baseline to 9 Months
Description: The Aggression Questionnaire (AQ) is a 34-item questionnaire that rates five types of aggression (physical aggression, verbal aggression, anger, hostility, and indirect aggression). Item responses ranged from 1-5, with 1=Not at all like me, 2=A little like me, 3=Somewhat like me, 4=Very much like me, 5=Completely like me. Higher scores indicate more aggression.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
score on a scale
  Baseline AQ Total | 2.02 (0.52) | 2.01 (0.52)
  3-month AQ Total | 2.09 (0.61) | 2.02 (0.61)
  9-month AQ Total | 2.03 (0.55) | 1.99 (0.6)
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.07 — 3-month follow-up between groups effect size of general aggression
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .01 — 9-month follow-up between groups effect size of general aggression

3. Primary Outcome: Change in Attitudes About Relationship Violence From Baseline to 9 Months
Description: Adolescent Relationship Violence Questionnaire (ARVQ) is a 22-item questionnaire is a composite measure developed to assess changes in knowledge, attitudes, and methods of dealing with relationship violence. Item responses ranged from 1-4 with 1=strongly agree, 2=agree, 3=disagree 4=strongly disagree. Higher scores indicate more favorable attitudes.
Time Frame: Baseline, 3 months, and 9 months
Population: COMPLETER ANALYSIS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
score on a scale
  Adolescent Baseline ARVQ | 3.01 (0.28) | 2.98 (0.30)
  Adolescent 3-month ARVQ | 3.03 (0.33) | 3.00 (0.34)
  Adolescent 9-months ARVQ | 3.10 (0.34) | 3.02 (0.34)
  Parent Baseline ARVQ | 3.43 (0.33) | 3.47 (0.29)
  Parent 3-month ARVQ | 3.45 (0.31) | 3.53 (0.30)
  Parent 9-month ARVQ | 3.44 (0.32) | 3.51 (0.31)
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .01 — 3-month follow-up between groups effect size of adolescent attitudes support aggression
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.17 — 9-month follow-up between groups effect size of adolescent attitudes support aggression
Statistical Analysis 3: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .19 — 3-month follow-up between groups effect size of parent attitudes support aggression
Statistical Analysis 4: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .20 — 9-month follow-up between groups effect size of parent attitudes support aggression

4. Secondary Outcome: Change in Emotion Regulation Skills From Baseline to 9 Months
Description: The Adolescent Self-Regulatory Inventory (ASRI) is a 33 item survey that measures adolescents' use of both functional and dysfunctional emotion regulation strategies. It produces two sub scales measuring short-term and long-term self-regulation. Item responses range from 1-5 with 1= Not at all true for me, 2= Rarely true for me, 3= True some of the time, 4= True most of the time, 5= Really true for me. Items were reverse coded so that higher scores indicate more use of emotion regulation behaviors.
Time Frame: Baseline, 3 months, and 9 months
Population: COMPLETER ANALYSIS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
score on a scale
  Baseline Short-Term Self-Regulation | 3.60 (0.65) | 3.63 (0.67)
  3-month Short-Term Self-Regulation | 3.55 (0.76) | 3.63 (0.71)
  9-month Short-Term Self-Regulation | 3.44 (0.80) | 3.71 (0.75)
  Baseline Long-Term Self-Regulation | 3.22 (0.57) | 3.23 (0.50)
  3-month Long-Term Self-Regulation | 3.24 (0.55) | 3.21 (0.52)
  9-month Long-Term Self-Regulation | 3.23 (0.51) | 3.33 (0.58)
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .09 — 3-month follow-up between groups effect size of adolescent short-term self-regulation
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .36 — 9-month follow-up between groups effect size of adolescent short-term self-regulation
Statistical Analysis 3: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.11 — 3-month follow-up between groups effect size of adolescent long-term self-regulation
Statistical Analysis 4: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .11 — 9-month follow-up between groups effect size of adolescent long-term self-regulation

5. Secondary Outcome: Change in Parent-Adolescent Communication From Baseline to 9 Months
Description: Parent Adolescent Communication Survey (PACS) is 20 item survey measuring quality of communication between adolescents and their parents. Adolescents will complete the measure in reference to the parent participating in the intervention with them. This is completed by parents and youth. This scale also produces two sub scales: The Open Family Communication Scale (OFCS) and The Problems in Family Communication Scale (PFCS). Item responses range from 1-5 with 1=Strongly disagree, 2=Moderately disagree, 3=Neither agree neither disagree, 4=Moderately agree, 5=Strongly agree. On the OFCS subscale, higher scores indicate more open communication. One the PFCS subscale, higher scores indicate fewer problems in family communication, thus higher scores on both subscales are favorable.
Time Frame: Baseline, 3 months, and 9 months
Population: COMPLETER ANALYSIS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
score on a scale
  Adolescent Baseline OFCS | 38.65 (8.08) | 37.65 (10.05)
  Adolescent 3-months OFCS | 36.65 (9.82) | 36.87 (10.18)
  Adolescent 9-month OFCS | 35.13 (9.96) | 35.16 (11.23)
  Adolescent Baseline PFCS | 34.39 (6.52) | 32.46 (7.23)
  Adolescent 3-month PFCS | 34.11 (7.40) | 31.98 (6.98)
  Adolescent 9-month PFCS | 33.60 (8.03) | 33.12 (7.69)
  Adolescent Baseline # of Relationship Topics | 3.24 (1.79) | 3.05 (2.14)
  Adolescent 3-month # of Relationship Topics | 1.88 (2.18) | 2.96 (2.43)
  Adolescent 9-month # of Relationship Topics | 1.80 (2.00) | 1.96 (2.05)
  Parent Baseline OFCS | 40.17 (6.98) | 39.33 (5.89)
  Parent 3-month OFCS | 40.18 (7.41) | 40.73 (6.06)
  Parent 9-month OFCS | 40.55 (6.71) | 40.16 (6.80)
  Parent Baseline PFCS | 37.35 (5.63) | 38.65 (5.68)
  Parent 3-month PFCS | 37.52 (5.58) | 39.25 (5.29)
  Parent 9-month PFCS | 38.06 (6.13) | 40.20 (5.05)
  Parent Baseline # of Relationship Topics | 4.32 (1.83) | 4.20 (1.79)
  Parent 3-month # of Relationship Topics | 3.36 (2.05) | 4.56 (1.65)
  Parent 9-month # of Relationship Topics | 3.70 (2.06) | 3.57 (1.89)
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .11 — 3-month follow-up between groups effect size of adolescent reported open family communication
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .06 — 9-month follow-up between groups effect size of adolescent reported open family communication
Statistical Analysis 3: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.15 — 3-month follow-up between groups effect size of adolescent reported problems in family communication
Statistical Analysis 4: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .06 — 9-month follow-up between groups effect size of adolescent reported problems in family communication
Statistical Analysis 5: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .62 — 3-month follow-up between groups effect size of adolescent reported number of relationship topics discussed
Statistical Analysis 6: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .13 — 9-month follow-up between groups effect size of adolescent reported number of relationship topics discussed
Statistical Analysis 7: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .15 — 3-month follow-up between groups effect size of parent reported open family communication
Statistical Analysis 8: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .01 — 9-month follow-up between groups effect size of parent reported open family communication
Statistical Analysis 9: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.15 — 3-month follow-up between groups effect size of parent reported problems in family communication
Statistical Analysis 10: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .25 — 9-month follow-up between groups effect size of parent reported problems in family communication
Statistical Analysis 11: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .66 — 3-month follow-up between groups effect size of parent reported number of relationship topics discussed
Statistical Analysis 12: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.10 — 9-month follow-up between groups effect size of parent reported number of relationship topics discussed

6. Secondary Outcome: Change in Emotion Regulation Skills Baseline to 9 Months
Description: The Emotion Regulation Behavioral Skills (ERBS) scale is comprised of 8 items rated on a scale of 1 "all the time" to 5 "never" and was specifically created for to detect the use of the specific affect management strategies taught in the Project STRONG intervention. Sample items include "How often did you…get away from whatever was causing your feeling? …talk to someone about whatever was causing your feeling?" Higher scores indicate greater use of emotion regulation skills.
Time Frame: Baseline, 3 months, 9 months
Population: COMPLETER ANALYSIS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
score on a scale
  Baseline ERBS | 2.04 (0.82) | 2.18 (0.82)
  3-month ERBS | 2.01 (0.83) | 2.18 (0.92)
  9-month ERBS | 1.86 (0.70) | 2.21 (0.91)
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .15 — 3-month follow-up between groups effect size of adolescent emotion-regulation
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .32 — 9-month follow-up between groups effect size of adolescent emotion-regulation

7. Secondary Outcome: Change in Distress Tolerance From Baseline to 9 Months
Description: The Behavioral Indicator of Resiliency to Distress (BIRD) is a 5-minute computerized distress tolerance task for adolescents. This measure generates a score of total time that adolescents persist on a frustrating task, which has been linked to distress tolerance. Scores are recorded in milliseconds (ms) with a maximum time participants can persist is 300 seconds (0-300 is the range). Higher score indicate longer persistence during the frustrating task.
Time Frame: Baseline, 3 months, 9 months
Population: COMPLETER ANALYSIS
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Waitlist Control | Project STRONG
Number analyzed (Participants) | 60 | 54
seconds
  Baseline BIRD | 256.68 (78.70) | 251.19 (78.05)
  3-month BIRD | 240.98 (80.06) | 230.66 (84.04)
  9-month BIRD | 227.17 (84.39) | 243.14 (78.35)
Statistical Analysis 1: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = -.11 — 3-month follow-up between groups effect size of adolescent distress tolerance
Statistical Analysis 2: Comparison: Waitlist Control vs Project STRONG; Test type: Superiority; Effect Size (d) = .23 — 9-month follow-up between groups effect size of adolescent distress tolerance

ADVERSE EVENTS:
Time Frame: 9 months
Description: Adverse events, as defined by clinicaltrials.gov, were monitored for Parents and Teens throughout the course of the trial
Groups:
- Waitlist Control: Parents-teen dyads enrolled in the study and randomized to the control condition wait until they complete their 3-month and 9-month follow-up surveys before completing the web-based program.
- Project STRONG: The web-based program consists of a number of games, activities, and didactic information that teens move through with their parent. Didactic information introduces teens and parents to specific emotion management, communication, and problem solving strategies as well as sexual health and healthy relationship information. Games and activities allow parent-teen dyads to practice and apply strategies to developmentally appropriate situations.
Arm/Group | Waitlist Control | Project STRONG
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/59

LIMITATIONS AND CAVEATS:
The primary limitation of this pilot Randomized Controlled Trial was the small sample size. A larger trial with more diverse group of families is needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03109184/Prot_SAP_000.pdf